CLINICAL TRIAL: NCT02646033
Title: Quantitative Rise in Intraocular Pressure in Steep Trendelenburg Position
Status: Completed | Type: Observational
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Dr. Nitesh Goel, Doctor, Consultant Anaesthesia, Rajiv Gandhi Cancer Institute & Research Center, India
Other Study IDs: RajivGCIRC
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Intraocular Pressure
Keywords: Intraocular Pressure, Trendelenburg position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- robotic surgery: all those patients aged 40 - 60 years undergoing robotic surgeries, who does not have any ophthalmic complains.

SUMMARY:
This study analyse the rise in Intraocular Pressure while patient is in surgery in head low position.

DETAILED DESCRIPTION:
Patient undergoing robotic surgeries requires steep trendelenburg position (upto 60 degrees) along with pneumoperitoneum. These both can cause a significant rise in intraocular pressure. Significant rise of pressure for prolonged period can cause post operative visual disturbances, which can be of medicolegal importance. Thus studying the quantitative rise and thus trend of intraocular pressure is first step in managing ophthalmic changes during robotic surgeries.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) status 1-3
* without any ophthalmic complains or interventions

Exclusion Criteria:

* lasix given during preoperative or intraoperative period
* cardiac patients who are on medications for stents or post Coronary Artery Bypass Graft (CABG)
* pre-existing glaucoma, eye surgeries, cataract or retinal vascular diseases, corneal diseases which may affect IOP measurement were excluded

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing robotic surgeries in steep trendelenburg position
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | 7-8 months
  change in pressure with the position during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nitesh Goel, MBBS,DA, DNB, Principal Investigator — Rajiv Gandhi Cancer Institute & Research Centre
Locations (1):
- Rajiv Gandhi Cancer Institute & Research Centre, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No